CLINICAL TRIAL: NCT01685918
Title: Safety and Effectiveness of Biological DMARDs in Elderly Patients With Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hanyang University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Sang-Cheol Bae, Professor, MD, PhD, MPH, Hanyang University
Other Study IDs: ederly_RA
Record Dates: First submitted 2012-09-12; First posted 2012-09-14 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; aged
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Study objectives

1. Comparison of drug persistency rates between elderly RA patients and young RA patients with biological DMARDs
2. Analysis of discontinuation reasons & influencing factors of drug discontinuation in elderly RA patients and young RA patients
3. Comparison of the occurrence of adverse events & treatment outcomes between elderly RA patients and young RA patients

DETAILED DESCRIPTION:
1. Retrospective study:

   We will collect data of Korean patients with RA retrospectively. Subjects will be extracted from medical records of RA patients who had treated with TNF inhibitor or are currently using TNF inhibitor. Patients who have received or are receiving biologic agents including infliximab, etanercept, adalimumab, rituximab from Dec.2000 to Dec.2010 will be enrolled.

   Data for this study which are sex, date of birth, previous and current medication, the results of laboratory test, disease activity of RA (DAS28ESR), comorbidity will be collected. Information of treatment, DAS28ESR, laboratory data and SAEs will be collected at baseline and predefined time points of follow-up (0, 3 month and recent follow-up data).

   During the first year of starting our study, we will focus to evaluate tolerability, the reason of discontinuation in elderly RA patients through this retrospective study. Tolerance could be analyzed by examining drug persistency of biologic DMARDs with the reason that led to drug interruption, and the drug persistency curves will be compared in the two groups. The length of time that patients remain on the drug therapy represents a useful measure of the treatment effectiveness and tolerability. The reason of discontinuation will be evaluate as descriptive analysis. And factors influenced on drug discontinuation in elderly RA patients and young RA patients using Cox-proportional analysis.
2. Prospectively study:

We will use the data of patients of Hanyang University Hospital for Rheumatic Diseases in web-based registry of RA patients with biologic DMARDs. Patients who start on receiving biologic agents including infliximab, etanercept, adalimumab, rituximab, abatacept will be enrolled. At registration, sex, date of birth, previous and current medication, the results of laboratory test, disease activity of RA (DAS28ESR), HAQ, comorbidity, socioeconomic status, etc. will be collected. Information of treatment, DAS28ESR, HAQ, laboratory data and SAEs, etc. will be collected at baseline and predefined time points of follow-up (0, 3 month and every 6 month). This prospective study will be progressed during three years.

We will focus the response of biologic DMARDs and the occurrence of adverse event in elderly RA patients in this prospective study. The response could be evaluated with the change of DAS28ESR and functional disability (HAQ). We will compare the response in elderly RA patients versus young RA patients, and evaluate the impact of old age on the response using multiple logistic regression model with adjust various confounding factors. The occurrence of adverse events during three years will be described in two groups

ELIGIBILITY:
Inclusion Criteria:

1. Retrospective study

   * Patients who satisfy the 1987 ACR classification criteria for RA
   * Patients with RA who have received or are receiving biologic agents including infliximab, etanercept, adalimumab, rituximab.
2. Prospective study

   * Patients who satisfy the 1987 ACR classification criteria for RA
   * Patients with RA who have received or are receiving biologic agents including infliximab, etanercept, adalimumab, rituximab, abatacept.

Exclusion Criteria:

1. Patients younger than eighteen
2. Patients enrolled in clinical trials
3. For the prospective study: Sex and Reproductive Status

   1. WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 10 weeks after the last dose of study drug.
   2. Women who are pregnant or breastfeeding.
   3. Women with a positive pregnancy test on enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Retrospective study: 425 patients with RA We will collect data of Korean patients with RA retrospectively. Subjects will be extracted from medical records of RA patients who had treated with biological DMARDs or are currently using biological DMARDs from Dec 2000 to Dec 2010.
  2. Prospectively study: 203 patients with RA We will use the web-based registry of RA patients with biologic DMARDs. This prospective study will be progressed during three years.
  We will compare the response in elderly RA patients versus young RA patients, and evaluate the impact of old age on the response. The occurrence of adverse events during three years will be described.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
drug(biologics) persistency rates | Patients who have received or are receiving biologic agents including infliximab, etanercept, adalimumab, rituximab from Dec.2000 to Dec.2010 will be enrolled.
  The tolerability in the two groups (elderly RA patients and young RA patients) will be estimated by drug persistency rates using the Kaplan-Meier method. Comparisons between the resultant curves will be made by log rank test.

SECONDARY OUTCOMES:
Treatement response (HAQ, DAS28) | Information of treatment, DAS28ESR, HAQ, laboratory data and SAEs, etc. will be collected at baseline and predefined time points of follow-up (0, 3 month and every 6 month). This prospective study will be progressed during three years.
  Treatments outcomes will be compared between two groups (elderly RA patients and young RA patients). The significance of differences in mean values of continuous variables will be assessed with Student's t-test. We will evaluate the impact of old age on the response using Cox proportional hazard analysis with adjust various confounding factors.

CONTACTS AND LOCATIONS:
Overall Officials: Sang-cheol Bae, Director, Principal Investigator — Hanyang University Hospital for Rheumatic Disease
Locations (1):
- Hanyang University Hospital for rheumatic disease, Seoul, Sung-dong Gu, South Korea